CLINICAL TRIAL: NCT00046189
Title: Cancer Risk in Xeroderma Pigmentosum Heterozygotes
Brief Title: Cancer Risk in Carriers of the Gene for Xeroderma Pigmentosum
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020313; 02-C-0313; NCT00049621 (obsolete NCT alias)
Record Dates: First submitted 2002-09-21; First posted 2002-09-23 (Estimated); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Xeroderma Pigmentosum; Basal Cell Carcinoma; Squamous Cell Carcinoma; Melanoma; Skin Cancer
Keywords: Sun Exposure; Xeroderma Pigmentosum; Skin Cancer; Family History; HETEROZYGOTE; Natural History; XP
MeSH Terms: conditions — Xeroderma Pigmentosum; Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Melanoma; Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Patients with XP
- 2: Family members from XP families with known DNA repair gene mutations

SUMMARY:
This study will determine if family members of patients with xeroderma pigmentosum (XP) have various abnormalities, including: skin abnormalities; nervous system abnormalities, such as hearing problems; skin, eye, or internal cancers, or other changes. XP is a rare inherited disease that involves an inability to repair damage to cell DNA (genetic material). It can affect several organ systems, including the skin, eye, nervous system, and bones. Patients have a more than thousand-fold increase in frequency in all major skin cancers.

Parents of patients with XP are carriers of the abnormal XP gene. Other family members may also be carriers of the abnormal XP gene. Carriers do not develop the disease themselves; symptoms develop only in children who have inherited the faulty gene from both parents. This study will try to clarify the genetic basis for XP and to understand the increased frequency of cancer in the disease.

XP patients who have been evaluated at the NIH Clinical Center and their relatives are eligible for this study. Newly diagnosed XP patients are also eligible. Spouses of relatives will also be included as control subjects.

Patients and their family members will undergo some or all of the following procedures:

* Parental permission to review the child s relevant medical records and pathology material from treatments or surgery for cancer or other related illnesses
* Medical history and physical examination, with particular attention to the skin and possible eye, hearing or neurological examinations
* Photographs to document skin and other physical findings
* Nuclear medicine scans to evaluate the brain and nervous system
* X-rays of the skull or other parts of the body
* Nervous system testing with an electroencephalogram (EEG), electroretinogram (ERG), electromyogram (EMG) or nerve conduction velocity measurement
* Collection of blood and skin samples for gene studies
* Establishment of cell lines from collected blood or tissues to study DNA repair, skin cancer, cancers related to XP, immune defects, and related studies.
* Biopsy (surgical removal of a small piece of tissue) of suspicious skin lesions for examination under a microscope
* Collection of a cheek cell sample, obtained by twirling a soft brush against the inside of the cheek
* Collection of a hair sample for microscopic examination and composition analysis
* Surgery to treat skin cancers or other lesions

DETAILED DESCRIPTION:
Xeroderma Pigmentosum (XP) is a rare, recessive disorder with a more than 1000-fold increase in the frequency of all major skin cancers in association with defective DNA repair. The risk of skin and other cancers among normal appearing XP heterozygote individuals has not been fully studied. We plan to study the family members from XP families with known DNA repair gene mutations to determine if heterozygote carriers of XP disease mutations are at an increased risk of developing cancer. For controls we will compare XP heterozygotes to their non-carrier blood relatives and spouses and to the Surveillance, Epidemiology and End Results (SEER) rates. For this purpose, blood, skin or buccal cells will be obtained from all available relatives for DNA or RNA mutation analysis. Cancer confirmation will be accomplished through review of pathology reports, medical records and death certificates. In addition, willing family members will be clinically examined to determine current cancer status. Individuals who are determined to be heterozygous carriers of XP DNA repair gene disease mutations in these families by mutation analysis or by pedigree will be compared to non-carrier relatives and spouses with respect to history of any type of cancer. We will also focus on skin cancer and cancer of the nervous system since the risks of these cancers are elevated among the XP homozygotes.

ELIGIBILITY:
* INCLUSION CRITERIA:

Members of the XP families where the proband has previously been evaluated at the Clinical Center or is newly diagnosed under other approved protocols (primarily 99-C-0099) are eligible to participate in this study. Families with XP patients of any age (excluding neonates), gender or race are eligible for this study.

* On referral, patients with XP and families of XP patients will be considered for inclusion in the study if the proband has clinical documentation of features of XP and laboratory determination of the DNA repair defect. All relatives of XP patients including spouses are eligible to participate. A spouse of a blood relative of a patient with xeroderma pigmentosum would also be eligible.
* Ability of patient or Legally Authorized Representative (LAR) to sign a written informed consent document

EXCLUSION CRITERIA:

-Inability or unwillingness to provide family history information or tissue (skin, blood, buccal cells or hair) for laboratory studies.

Ages: 1 Month to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with XP families where the proband has previously been evaluated at the Clinical Center or is newly diagnosed
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2003-04-07 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Determine increased risk of developing cancer | Annual
  risk of any type of cancer, skin cancer and cancers of the nervous system are compared in the relatives who are heterozygotes for the XP mutations and relatives who do not carry the XP mutations by calculating the odds ratios

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H Kraemer, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-C-0313.html